CLINICAL TRIAL: NCT02503956
Title: The Efficacy of Punctal Dilatation With Insertion of Perforated Punctal Plugs for the Management of Acquired Punctal Stenosis Due to Allergic Conjunctivitis
Brief Title: Perforated Punctal Plugs for Treatment of Papillary Conjunctivitis in Otherwise Healthy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Alpha Net Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0557-14-RMC
Record Dates: First submitted 2015-06-24; First posted 2015-07-21 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-02

CONDITIONS: Epiphora; Conjunctivitis
MeSH Terms: conditions — Lacrimal Apparatus Diseases; Conjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treated group (Experimental): Patients treated with perforated punctal plugs
  Interventions: Device: Perforated Punctal plugs
- Comparison group (Active Comparator): Comparison group treated with standard of care - Lacrimal intubation with Crawford lacrimal tube
  Interventions: Procedure: Crawford tube insertion; Device: Crawford lacrimal tube

INTERVENTIONS:
Device: Perforated Punctal plugs — Perforated punctal plugs
  Arms: Treated group
Procedure: Crawford tube insertion
  Arms: Comparison group
Device: Crawford lacrimal tube
  Arms: Comparison group

SUMMARY:
Assessing efficacy of punctal dilatation with insertion of perforated punctal plugs for the management of acquired punctal stenosis due to allergic conjunctivitis in otherwise healthy patients.

DETAILED DESCRIPTION:
The efficacy of punctal dilatation with insertion of perforated punctal plugs for the management of acquired punctal stenosis due to allergic conjunctivitis.

Acquired punctal stenosis is a condition in which the external opening of the lacrimal canaliculus is narrowed or occluded due to chronic inflammation and fibrosis. This condition is a rare cause of symptomatic epiphora, but its incidence may be higher in patients with chronic blepharitis, in those treated with various topical medications, including antihypertensive agents, and especially in patients treated with taxanes for cancer.

The incidence of punctal stenosis is still unknown, with reported rates ranging from 8% to 54.3%, depending on setting, demographics, and probably interob¬server variability. Nevertheless, the literature suggests that this pathology should be given special consideration while assessing the tearing patient, because it may involve an easier surgical solution than in patients with obstruction in the more distal lacrimal system.

Recently many oculoplastic surgeons encounter young patients (usually females) with punctual stenosis and signs of allergic conjunctivitis but no reflex tearing. In these cases, treatment for allergic conjunctivitis does not improve tearing. Treatment with punctoplasty of mini- Monoka stents improve their condition for the short term. However, many patients experience recurrence of epiphora in the long term.

There are no uniform clinical guidelines for treatment of the disease. A few methods are currently used in the management of punctal stenosis. The most common in use are punctoplasty or intubation with minimonoka stents. Substantial experience with these minor surgical snip procedures would suggest giving preference to their utilization in the treatment of the disease in our clinics.

The simplest method involves the use of perforated punctal plugs, a reversible simple procedure that can be applied in an office setting. Silicon perforated plugs are inserted after punctual dilatation under topical anesthesia to the lacrimal punctum in order to maintain a patent tear drain into the nasolacrimal sac. The procedure is simple and usually pain free. After the procedure topical steroids and antibiotics are prescribed for one week. Plugs are extracted after a two month period in the outpatient clinic.

Unfortunately, evidence for the efficacy of the procedure for acquired punctual stenosis is scarce. One retrospective series of 44 eyes from 26 patients treated with dilation and the placement of a perforated punctal plug for acquired punctal stenosis, the success rate was 84.1% (37 of 44 eyes) for cessation of epiphora. The plugs were extracted after 2 months. Most cases had partial punctal stenosis. Associated eyelid laxity was detected in 14 eyes, and eight of them underwent a lateral tarsal strip procedure prior to plug implantation. The mean follow-up period was 19 months. Failures were due to either restenosis or horizontal eyelid laxity.

Another study evaluated the use of perforated punctual plugs in patients with acquired punctual stenosis, 20 patients in total. This study showed 85% successes rate in total. Patients where the procedure failed were usually older and were likely to have blepharitis.

Although perforated punctal plugs are an attractive non¬surgical tool in the management of acquired punctal stenosis, the long-term results of the procedure and its role in treating punctal stenosis requires and prospective larger clinical trials.

Study design We intend to perform a prospective clinical trial to assess the efficacy of perforated punctual plugs in treating acquired punctual stenosis. Since patients were previously assigned to treatment by a Crawford tube insertion, this patient group will act as the comparison group for this study.

Adult, consenting patients will be recruited from the ophthalmology outpatient clinics in Rabin Medical Center. Punctal plugs will be inserted in the outpatient clinics for duration of two months.

Plug insertion will be performed under topical anesthesia after careful dilation of the lacrimal punctum. Patients will be prescribed topical steroids and antibiotic for a one week period following plug insertion procedure. Punctal plugs will be removed after two months treatment period. Follow up time is intended for two years to asses both short term and long term efficacy.

Records for patients who underwent Crawford tube insertion due to allergic conjunctivitis will be anonymously collected from Rabin Medical Centers' database. The collected data will be analyzed and used a comparison group for the study.

ELIGIBILITY:
Inclusion Criteria

* Patients suffering from acquired punctual stenosis due to chronic allergic conjunctivitis.
* 18 - 100 Years old
* Able to sign an informed consent and agree to participate Exclusion Criteria
* Previous manipulation of lacrimal ducts of punctum
* Patients unable to follow study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07-22 (Actual); Study Completion 2016-07-22 (Actual)

PRIMARY OUTCOMES:
Epiphoric state | 3 Months
  Patient follow up after punctal plug removal, this is a dichotomic measure of yes/no question - weather of not the patient still suffers from tearing after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Itay Gabbay, MD, Principal Investigator — Physician
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Result] Ali MJ, Mishra DK, Baig F, Lakshman M, Naik MN. Punctal stenosis: histopathology, immunology, and electron microscopic features-a step toward unraveling the mysterious etiopathogenesis. Ophthalmic Plast Reconstr Surg. 2015 Mar-Apr;31(2):98-102. doi: 10.1097/IOP.0000000000000204. PMID 24892278
- [Result] Soiberman U, Kakizaki H, Selva D, Leibovitch I. Punctal stenosis: definition, diagnosis, and treatment. Clin Ophthalmol. 2012;6:1011-8. doi: 10.2147/OPTH.S31904. Epub 2012 Jul 3. PMID 22848141
- [Result] Konuk O, Urgancioglu B, Unal M. Long-term success rate of perforated punctal plugs in the management of acquired punctal stenosis. Ophthalmic Plast Reconstr Surg. 2008 Sep-Oct;24(5):399-402. doi: 10.1097/IOP.0b013e318185a9ca. PMID 18806663
- [Result] Mathew RG, Olver JM. Mini-monoka made easy: a simple technique for mini-monoka insertion in acquired punctal stenosis. Ophthalmic Plast Reconstr Surg. 2011 Jul-Aug;27(4):293-4. doi: 10.1097/IOP.0b013e31820ccfaf. PMID 21386741
- [Result] Hussain RN, Kanani H, McMullan T. Use of mini-monoka stents for punctal/canalicular stenosis. Br J Ophthalmol. 2012 May;96(5):671-3. doi: 10.1136/bjophthalmol-2011-300670. Epub 2012 Jan 12. PMID 22241928
- [Result] Chang M, Ahn SE, Baek S. The effect of perforated punctal plugs in the management of acquired punctal stenosis. J Craniofac Surg. 2013 Sep;24(5):1628-30. doi: 10.1097/SCS.0b013e318292c68b. PMID 24036740